CLINICAL TRIAL: NCT06892366
Title: Effects of Home-Based Aerobic and Resistance Exercise on Oxygen Consumption, Muscle Function, Frailty, Quality of Life, and Health-Related Lifestyle in Chronic Liver Disease
Brief Title: Impact of Home-Based Aerobic and Resistance Training in Chronic Liver Disease: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Bilge Taskin Gurel, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BTG
Record Dates: First submitted 2025-01-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Liver Disease and Cirrhosis
Keywords: end-stage liver disease; exercise; sarcopenia
MeSH Terms: conditions — Fibrosis; End Stage Liver Disease; Motor Activity; Sarcopenia | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Exercise (AE) Group (Experimental): Participants in this group performed moderate-intensity aerobic exercises, primarily walking, three non-consecutive days per week for eight weeks. Exercise intensity was set at 40-60% of peak VO2 or based on perceived exertion (Borg 4-6) for those on beta-blockers. Sessions were monitored via video conferencing, and participants used smart wristbands for heart rate tracking.
  Interventions: Behavioral: Home-Based Aerobic Exercise Program
- Aerobic and Resistance Exercise (ARE) Group (Experimental): Participants in this group performed a combination of aerobic and resistance exercises. Aerobic sessions followed the same protocol as the AE group (3 days/week). Resistance exercises were performed 2 additional days per week using elastic resistance bands calibrated to 40-50% of 1RM. Each resistance session included 3 sets of 10 repetitions for major muscle groups. All sessions were conducted and monitored remotely.
  Interventions: Behavioral: Home-Based Aerobic and Resistance Exercise (ARE) Group
- Control Group (No Intervention): This group does not receive a structured exercise intervention. While they are monitored for daily step counts and encouraged to stay active, there is no specific intervention implemented.

INTERVENTIONS:
Behavioral: Home-Based Aerobic Exercise Program — Aerobic Exercise (AE) Group This intervention consists of a home-based aerobic exercise program emphasizing moderate-intensity walking, tailored to 40-60% of peak VO2 or Borg Scale 4-6 for those on beta blockers. Distinctive features include real-time session supervision via video conferencing and heart rate monitoring with a smart wristband. This approach ensures remote guidance, personalized intensity, and participant safety throughout the 8-week program.
  Arms: Aerobic Exercise (AE) Group
Behavioral: Home-Based Aerobic and Resistance Exercise (ARE) Group — Participants engaged in a combined home-based aerobic and resistance exercise program. Aerobic sessions followed the same protocol as the AE group (3 days/week). Resistance training was performed 2 additional days per week using elastic resistance bands set at 40-50% of one-repetition maximum (1RM). Resistance exercises targeted major muscle groups, with each session consisting of 3 sets of 10 repetitions, and 1-3 minutes of rest between sets. All sessions were monitored and supervised remotely.
  Arms: Aerobic and Resistance Exercise (ARE) Group

SUMMARY:
The goal of this clinical trial is to evaluate whether home-based exercise interventions, including aerobic exercise (AE) and a combination of aerobic and resistance exercise (ARE), can improve physical and health-related outcomes in patients with chronic liver disease (CLD). The primary population includes adult patients with CLD experiencing complications such as sarcopenia, malnutrition, and fatigue.

The main questions it aims to answer are:

Does home-based ARE improve oxygen consumption, muscle strength, and physical frailty more effectively than AE or no exercise? Can home-based exercise reduce fatigue and improve quality of life and health-related behaviors?

Researchers will compare the outcomes of three groups:

Home-based AE group Home-based ARE group Control group (physical activity counselling)

Participants will:

Perform an 8-week home-based exercise program based on their group allocation (either AE or ARE).

Undergo evaluations before and after the intervention, including:

Oxygen consumption (via cardiopulmonary exercise testing) Muscle strength (using a hand dynamometer and respiratory muscle strength tests) Body composition (via bioelectrical impedance analysis and skinfold thickness measurements) Quadriceps muscle thickness and cross-sectional area (using muscle ultrasound) Muscle oxygenation Fatigue levels (using the Fatigue Severity Scale) Physical frailty (using the Liver Frailty Index) Quality of life (using the Chronic Liver Disease Questionnaire) Health-related lifestyle behaviors (using the Health-Promoting Lifestyle Profile II)

DETAILED DESCRIPTION:
This randomized controlled trial was designed to evaluate the effects of an 8-week home-based exercise program on physical and health-related outcomes in patients with Chronic Liver Disease (CLD). The study included three groups: Aerobic Exercise (AE), Aerobic and Resistance Exercise (ARE), and a control group. Below are the details of the interventions and measurement techniques utilized in the study.

Study Groups and Interventions

1. Aerobic Exercise (AE) Group:

   Exercise Protocol: Participants engaged in moderate-intensity walking exercises three non-consecutive days per week. The intensity was set at 40-60% of peak VO2 (measured by cardiopulmonary exercise testing), or based on the perceived exertion scale (Borg 4-6) for those on beta-blockers.

   Session Structure:
   * 5 minutes warm-up: Stretching or light walking.
   * 20 minutes aerobic walking at target intensity.
   * 5 minutes cool-down: Stretching or light walking.

   Monitoring and Equipment: Heart rate monitoring was performed using Mi Smart Band 4. Sessions were conducted via video conferencing through WhatsApp, and pre-, during, and post-exercise feedback was recorded regarding heart rate, fatigue, and dyspnea.

   Safety Measures: Participants exercised in a safe indoor space cleared of obstacles, using appropriate footwear.
2. Aerobic and Resistance Exercise (ARE) Group:

   Exercise Protocol: Participants followed a combined regimen:

   Aerobic exercises (3 days/week) were conducted following the AE protocol. Resistance training (2 days/week) was performed with elastic resistance bands (TheraBand) set at 40-50% of 1RM.

   Resistance Training Exercises:
   * Targeted major muscle groups.
   * Each exercise involved 3 sets of 10 repetitions, with 1-3 minutes of rest between sets.
   * Resistance exercises were demonstrated and practiced during an initial session to ensure adherence.
   * Monitoring and Safety: Heart rate monitoring, perceived fatigue, and dyspnea were recorded before and after each session.
3. Control Group:

Participants received general guidance on physical activity benefits and were given Mi Smart Band 4 for activity monitoring.

Weekly phone calls were conducted to encourage increased step counts. Step counts were recorded during the first and eighth weeks for comparison.

Measurements and Assessments

Oxygen Consumption:

Measured using Cardiopulmonary Exercise Testing (CPET) on a treadmill (COSMED, Quark RMR) with the Modified Bruce Protocol. Peak VO2 and anaerobic thresholds were recorded, along with parameters such as ventilatory efficiency, heart rate, and metabolic equivalents.

Muscle Oxygenation:

Measured during CPET using near-infrared spectroscopy (NIRS) (Moxy, Fortiori Design LLC). Parameters included SmO2 and total hemoglobin changes (THb).

Peripheral Muscle Strength:

Assessed using a digital hand dynamometer (LaFayette Instrument Company) and isometric contractions. Strength of various muscle groups (e.g., quadriceps, hamstrings, shoulder abductors) was evaluated using standardized positions.

Respiratory Muscle Strength:

Maximal inspiratory (MIP) and expiratory pressures (MEP) were measured using a portable mouth pressure device (Micro RPM). Results were recorded in cmH2O and compared to age- and gender-specific predicted values.

Body Composition:

Measured using Bioelectrical Impedance Analysis (BIA) (Bodystat QuadScan 4000). Parameters included body fat percentage, lean mass, and phase angle. Skinfold measurements were performed using a caliper, and quadriceps muscle thickness and cross-sectional area were evaluated using ultrasound.

Frailty:

Evaluated using the Liver Frailty Index (LFI), which includes grip strength, sit-to-stand time, and balance tests. Scores classified participants as robust, pre-frail, or frail.

Physical Activity Levels:

Assessed using the International Physical Activity Questionnaire-Short Form (IPAQ). Scores were calculated in MET-min/week and classified as inactive, minimally active, or sufficiently active.

Fatigue:

Measured using the Fatigue Severity Scale (FSS), with responses recorded via an online form before and after the intervention.

Quality of Life:

Evaluated using the Chronic Liver Disease Questionnaire (CLDQ), addressing abdominal symptoms, fatigue, systemic symptoms, activity, emotional functioning, and anxiety.

Health-Related Lifestyle Behaviors:

Assessed using the Health-Promoting Lifestyle Profile II (HPLP-II), covering six domains: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.

Statistical Analysis Data were analyzed using descriptive and inferential statistics. Continuous variables were expressed as mean ± SD or median (min-max), while categorical variables were summarized as frequencies and percentages.

Dependent group comparisons: Paired t-tests or Wilcoxon Signed Rank tests were applied.

Independent group comparisons: ANOVA or Kruskal-Wallis tests, followed by post hoc tests (Tukey HSD or Mann-Whitney U).

A p-value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being followed up for chronic liver disease or listed on the liver transplant waiting list at the Hacettepe University Department of Internal Medicine, Division of Gastroenterology.
* Owning and being able to use a smartphone.
* Aged between 18 and 70 years.
* Receiving primary prophylactic treatment for gastroesophageal varices.
* Willingness to participate in the study.

Exclusion Criteria:

* Inability to own or use a smartphone.
* Participation in an exercise training program within the last year.
* Previous liver transplantation.
* High-risk varices without beta-blocker treatment.
* Presence of persistent hepatic encephalopathy.
* Hepatic hydrothorax.
* Pulmonary vascular complications of portal hypertension.
* Chronic renal failure requiring dialysis.
* Hemoglobin level below 10 g/dL.
* Creatinine level above 2 mg/dL.
* Human Immunodeficiency Virus (HIV) infection.
* Presence of hepatocellular carcinoma (HCC).
* Recent acute myocardial infarction.
* Uncontrolled arrhythmias causing symptomatic hemodynamic instability.
* Contraindications to maximal exercise testing.
* Physical or orthopedic conditions preventing home-based exercise training.
* Lack of willingness to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Peak Oxygen Consumption (VO₂ Max) | Baseline and at 8 weeks.
  Peak oxygen consumption (VO₂ Max) was measured using a Cardiopulmonary Exercise Test (CPET) conducted on a treadmill following the Modified Bruce Protocol. Ventilatory parameters were recorded breath-by-breath using a calibrated metabolic device (COSMED, Quark RMR, Rome, Italy) with an airtight face mask. The primary outcome was peak VO₂ (ml/min).
Relative Oxygen Consumption (VO₂/kg) | Baseline and at 8 weeks.
  Relative oxygen consumption (VO₂/kg) was measured as part of the Cardiopulmonary Exercise Test (CPET). The outcome was reported as VO₂/kg (ml/kg/min).
Anaerobic Threshold VO₂ | Baseline and at 8 weeks.
  The anaerobic threshold was determined using ventilatory parameters recorded during the Cardiopulmonary Exercise Test (CPET). The outcome was reported as VO₂ at the anaerobic threshold (ml/min).
Muscle Oxygenation (SmO₂) | Baseline and at 8 weeks.
  Muscle oxygenation (SmO₂) was measured during the Cardiopulmonary Exercise Test (CPET) using a near-infrared spectroscopy (NIRS) monitor (Moxy, Fortiori Design LLC, Minnesota, USA). The NIRS sensor was placed on the dominant leg's vastus lateralis muscle, positioned between the lateral epicondyle of the femur and the greater trochanter. SmO₂ values were recorded at rest (pre-test), at the end of CPET, and during recovery. The final 30 seconds of data were averaged for analysis at each stage. The reported outcome was the minimum SmO₂ value (%).
Change in Muscle Oxygenation During Exercise (ΔSmO₂) | Baseline and at 8 weeks.
  The change in muscle oxygenation (ΔSmO₂) was calculated as the difference between SmO₂ at rest (pre-test) and SmO₂ at peak exercise. The reported outcome was ΔSmO₂ (%).
Muscle Oxygenation During Recovery | Baseline and at 8 weeks.
  Recovery SmO₂ was measured as the SmO₂ value recorded 1 minute after exercise cessation. The reported outcome was recovery SmO₂ (%).
Total Hemoglobin (THb) | Baseline and at 8 weeks.
  Total hemoglobin (THb) was measured using near-infrared spectroscopy (NIRS) during CPET. THb values were recorded at rest, at peak exercise, and during recovery. The final 30 seconds of data were averaged at each stage. The reported outcome was the peak THb value (g/dL).
Peripheral muscle strength | Baseline and at 8 weeks.
  Peripheral muscle strength was measured using a digital hand dynamometer (LaFayette Instrument Company, Lafayette, Indiana, USA). The device recorded force in kilograms (kg), Newtons, and pounds. Participants were instructed to perform maximum isometric contractions during testing. Measurements were conducted for various muscle groups in standardized positions, including quadriceps, hamstrings, hip extensors, hip flexors, shoulder abductors, shoulder flexors, and scapular adductors. The dynamometer was positioned appropriately for each muscle group, such as 1-2 cm above the malleoli for knee extensors or on the posterior thigh proximal to the knee for hip extensors. Results were recorded in kilograms and analyzed for strength comparison across time points.
Respiratory muscle strength | Baseline and at 8 weeks.
  Respiratory muscle strength was assessed indirectly by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) using a portable mouth pressure device (Micro RPM, Care Fusion, Rochester, UK). Results were recorded in cmH2O. MIP was measured from residual lung volume, requiring participants to perform maximum inspiratory effort against a closed airway for 1-3 seconds. MEP was measured from total lung capacity, requiring maximum expiratory effort for 1-3 seconds. The highest value among three attempts with less than 10% variability was recorded. MIP and MEP values were expressed as percentages of age- and gender-predicted reference values at baseline and after the intervention.
Fat Mass | Baseline and at 8 weeks.
  Fat mass was measured using Bioelectrical Impedance Analysis (BIA) (Bodystat QuadScan 4000, Bodystat Ltd., Douglas, Isle of Man, UK). The reported outcome was fat mass (kg).
Lean Body Mass | Baseline and at 8 weeks.
  Lean body mass was assessed using Bioelectrical Impedance Analysis (BIA). The reported outcome was lean body mass (kg).
Total Body Water | Baseline and at 8 weeks.
  Total body water was measured as part of Bioelectrical Impedance Analysis (BIA). The reported outcome was total body water (liters).
Intracellular and Extracellular Fluid | Baseline and at 8 weeks.
  Intracellular and extracellular fluid were evaluated using Bioelectrical Impedance Analysis (BIA). The reported outcomes were intracellular fluid (liters) and extracellular fluid (liters).
Phase Angle | Baseline and at 8 weeks.
  Phase angle, a marker of cell membrane integrity and general health, was measured using Bioelectrical Impedance Analysis (BIA). The reported outcome was phase angle (degrees).
Rectus Femoris Muscle Thickness | Baseline and at 8 weeks.
  The thickness of the rectus femoris muscle was measured using ultrasound imaging (Logiq 200 Pro Ultrasound Device, General Electric, Chicago, Illinois, USA). The ultrasound transducer was placed perpendicular to the long axis of the femur, at a location two-thirds of the distance between the anterior superior iliac spine and the patella. Minimal pressure was applied to avoid compression of the muscle tissue during imaging. The reported outcome was rectus femoris muscle thickness (cm).
Rectus Femoris Cross-Sectional Area | Baseline and at 8 weeks.
  The cross-sectional area of the rectus femoris muscle was measured using ultrasound imaging. The transducer placement and imaging procedure were standardized to ensure consistent measurements. The reported outcome was rectus femoris cross-sectional area (cm²).
Physical Frailty (Liver Frailty Index) | Baseline and at 8 weeks.
  Physical frailty was assessed using the Liver Frailty Index (LFI), calculated with the following formula:
  LFI Score = (-0.030 x grip strength) + (-2.529 x sit-to-stand time) + (-0.040 x balance time) + 6.
  LFI includes:
  Grip Strength: Measured with a hand dynamometer in kilograms (kg). Sit-to-Stand Test: Time (seconds) to complete five sit-to-stand repetitions without hand support.
  Balance Test: Total time (seconds) maintaining feet-together, semi-tandem, and tandem stances (maximum 30 seconds).

SECONDARY OUTCOMES:
Physical Activity Level (IPAQ) | Baseline and at 8 weeks.
  Physical activity levels were assessed using the International Physical Activity Questionnaire-Short Form (IPAQ), validated in Turkish. The questionnaire includes seven items evaluating time spent sitting, walking, and performing moderate and vigorous physical activities over the past seven days. Activities performed for at least 10 continuous minutes were considered. MET-min/week scores were calculated by multiplying activity duration (minutes), frequency (days), and MET values (walking: 3.3 MET, moderate: 4.0 MET, vigorous: 8.0 MET). Total physical activity was classified as inactive, minimally active, or sufficiently active based on IPAQ scoring.
Quality of Life (Chronic Liver Disease Questionnaire - CLDQ) | Baseline and at 8 weeks.
  Quality of life was assessed using the Chronic Liver Disease Questionnaire (CLDQ), validated in Turkish. The CLDQ comprises six subdomains (abdominal symptoms, fatigue, systemic symptoms, activity, emotional function, and worry) and a total of 29 items. Each item is rated on a 7-point Likert scale, ranging from 1 ("always") to 7 ("never"). Higher total scores indicate better quality of life. Participants were asked to evaluate issues experienced in the past two weeks. The questionnaire was administered via an online platform (Google Forms) before and after the intervention.
Health-Promoting Lifestyle Behaviors (HPLP-II) | Baseline and at 8 weeks.
  Health-promoting lifestyle behaviors were assessed using the Health-Promoting Lifestyle Profile II (HPLP-II), validated in Turkish. The HPLP-II evaluates health-related behaviors across six subdomains: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management. The scale consists of 52 items rated on a 4-point Likert scale (1 = "never," 2 = "sometimes," 3 = "often," 4 = "always"), with higher scores indicating better health-promoting behaviors. The questionnaire was administered online via Google Forms before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar Yağlı, Prof, Study Director — Hacettepe University Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in any publication will be shared upon reasonable request. Data are securely stored at Hacettepe University and will be made available to researchers who provide a methodologically sound proposal, following applicable regulations and ethical guidelines. Access to data will be granted only for research purposes that align with the goals of this study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The individual participant data (IPD) will become available starting 6 months after the publication of the study's summary data or main results. The data will remain accessible for a period of 5 years following the initial availability date. Requests for access can be made during this time frame, subject to approval and adherence to institutional guidelines and ethical standards.
Access Criteria: Individual participant data (IPD) and supporting information will be shared with researchers who provide a methodologically sound proposal for scientific analyses that align with the objectives of this study. Requests will be reviewed by an institutional review committee at Hacettepe University to ensure compliance with ethical standards and data protection regulations. Approved researchers will be required to sign a data use agreement outlining conditions for use, storage, and confidentiality. Data will be shared securely through encrypted digital platforms.